CLINICAL TRIAL: NCT00004108
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Hepatocellular Carcinoma
Brief Title: DX-8951f in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067329; DAIICHI-8951A-PRT016; MDA-ID-99145; MSKCC-99058; UCHSC-00891
Record Dates: First submitted 1999-12-10; First posted 2004-04-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Liver Cancer
Keywords: localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating patients who have liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antitumor activity of DX-8951f in terms of antitumor response, response duration, and survival in patients with hepatocellular carcinoma. II. Assess the quantitative and qualitative toxicities of this treatment regimen in this patient population. III. Evaluate the pharmacokinetics of DX-8951 in plasma.

OUTLINE: Patients receive DX-8951f IV over 30 minutes daily for 5 days. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed hepatocellular carcinoma with or without evidence of unresectable extrahepatic metastasis Previously untreated disease OR Progressive disease after first line chemotherapy Bidimensionally measurable disease by CT scan, chest x-ray, or MRI of the abdomen No brain metastases

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 80,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL Albumin at least 2.8 g/dL SGOT/SGPT no greater than 5 times upper limit of normal (ULN) PT/INR no greater than 1.5 times ULN if not on coumadin therapy Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within the past 6 months Other: No concurrent serious infection No other life threatening illness No overt psychosis or mental disability that would preclude informed consent No other malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception 1 month prior to and during the study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No prior camptothecin analogues No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: No other concurrent anticancer therapy At least 4 weeks since prior investigational drugs (including analgesics or antiemetics) No other investigational drugs during or within 28 days after final dose of study drug

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Denver, Colorado
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas